CLINICAL TRIAL: NCT05327452
Title: Testing Home-based Exercise Strategies to Improve Exercise Participation and Cardiovascular Health in Underserved Minority Patients With Cancer Undergoing Chemotherapy: the THRIVE Study
Brief Title: Testing Home-based Exercise Strategies in Underserved Minority Cancer Patients Undergoing Chemotherapy: the THRIVE Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-559; 2U54CA156732-11 (NIH)
Record Dates: First submitted 2022-03-11; First posted 2022-04-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Colorectal Cancer; Prostate Cancer
Keywords: Breast Cancer; Colorectal Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised aerobic and resistance exercise (SUP) (Experimental): Participants will be randomly assigned to receive 3x weekly at home, virtually supervised aerobic and resistance exercise sessions with a certified exercise trainer for 16 weeks.
  Participants will also have a baseline test, mid intervention cardiovascular and strength tests and one postintervention and one follow up visit.
  Interventions: Behavioral: Supervised Home-Based Exercise
- Unsupervised aerobic and resistance exercise (UNSUP) (Experimental): Participants will be randomly assigned to receive 3x weekly at home, unsupervised aerobic and resistance exercise sessions with a 1x weekly telehealth call with a certified exercise trainer for 16 weeks.
  Participants will also have a baseline test, mid intervention cardiovascular and strength tests and one postintervention and one follow up visit.
  Interventions: Behavioral: Unsupervised Home-Based Exercise
- Attention Control (AC) (Active Comparator): Participants will be randomly assigned to receive 3x weekly at home stretching exercise for 16 weeks.
  Participants will also have a baseline test, mid intervention cardiovascular and strength tests and one postintervention and one follow up visit.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Supervised Home-Based Exercise — Online supervised aerobic and resistance exercise
  Arms: Supervised aerobic and resistance exercise (SUP)
Behavioral: Unsupervised Home-Based Exercise — Unsupervised aerobic and resistance exercise (UNSUP)
  Arms: Unsupervised aerobic and resistance exercise (UNSUP)
Behavioral: Attention Control — Stretching Program
  Arms: Attention Control (AC)

SUMMARY:
The purpose of this research is to determine whether a 16 week, home-based, aerobic and resistance exercise intervention will increase physical activity levels in Black and Hispanic breast, colorectal, or prostate cancer patients.

The names of the study interventions involved in this study are:

* Supervised aerobic and resistance exercise (SUP) - virtually supervised 16- week aerobic and resistance exercise performed at home via Zoom.
* Unsupervised aerobic and resistance exercise (UNSUP) - home-based 16- week aerobic and resistance exercise.
* Attention control (AC) - 16-week home-based stretching.

DETAILED DESCRIPTION:
This is a randomized control trial of Black and Hispanic patients who have been newly diagnosed with breast, colorectal, or prostate cancer and are being prescribed chemotherapy to determine the effects of home-based exercise on levels of physical activity. It will also evaluate the impact of home-based exercise on cardiovascular (heart health) risk factors.

The research study procedures include: screening for eligibility and study treatment including evaluations of body composition, blood tests, fitness and strength assessments, and surveys at study entry and follow-up visits.

Participants in this study will be randomly assigned to one of three groups: 1) Supervised aerobic and resistance exercise (SUP), 2) Unsupervised aerobic and resistance exercise (UNSUP), or 3) Attention control (AC).

Participation is expected to last for 8 months.

It is expected that about 135 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old; children under the age of 18 will be excluded due to rarity of disease
* Newly diagnosed with stage I-III breast, colorectal or prostate cancer
* Self-identify as Hispanic or Black
* Are within 4 weeks of initiating chemotherapy
* Overweight or obese (BMI >25kg/m2 or body fat percent >30)
* Physician's clearance to participate in moderate-vigorous intensity exercise
* Speak English or Spanish
* Engaging in less than 90 minutes of moderate-or-vigorous physical activity per week
* Willing to travel to Dana-Farber Cancer Institute for necessary data collection
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pre-existing musculoskeletal or cardiorespiratory conditions
* Patients should not have any uncontrolled illness including ongoing or active infection, uncontrolled diabetes, hypertension, or thyroid disease
* Patients with other active malignancies
* Patients with metastatic disease
* Participate in more than 90 minutes of structured exercise/week
* Unable to travel to Dana-Farber Cancer Institute for necessary data collection
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Activity Participation | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Changes from baseline in physical activity participation measured by Godin Leisure-Time Exercise Questionnaire.

SECONDARY OUTCOMES:
Biomarkers for Cardiovascular and Metabolic Health - insulin | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Fasting blood will be drawn from the antecubital vein by a trained phlebotomist. Insulin will be measured.
Blood Pressure | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Blood pressure will be assessed using an automated blood pressure cuff to measure both systolic and diastolic blood pressure.
Body Composition | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Body composition (lean mass and fat mass) will be assessed via bioelectrical impedance using a validated scale.
Cardiopulmonary Fitness | Evaluated at week 1 for baseline, week 9 for mid-point, week 16 for post-intervention assessment, and week 32 for follow-up
  Cardiopulmonary fitness will be measured by a submaximal graded exercise cycling test.
Physical Fitness | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Physical Fitness will be measured by the short physical performance battery (SPPB).
Cardiorespiratory Fitness | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Cardiorespiratory fitness will be assessed by the 6-minute walk test.
Muscular Strength | Evaluated at week 1 for baseline, week 9 for mid-point, week 16 for post-intervention assessment, and week 32 for follow-up
  Muscular strength will be assessed with a 10 repetition maximum test.
Patient Reported Outcomes - Quality of Life | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Quality of life will be assessed by EORTC QLQ C-30.
Patient Reported Outcomes - Health-related domains | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Health-related domains of patient reported outcomes will be assessed by PROMIS-29 Profile v2.1.
Patient Reported Outcomes - Sleep | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Quality of life will be assessed by the Pittsburg Sleep Quality Index (PSQI).
Patient Reported Outcomes - Symptoms | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Symptomatic toxicities will be assessed by PRO-CTCAE.
Dietary Assessment | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Dietary recall will be used to assess recent dietary patterns for two weekdays and one weekend day using NutriBase 11.
Acceptability of Intervention Questionnaire Ratings | Evaluated at months 2 and 4
  Intervention acceptability and feasibility will be assessed via Acceptability of Intervention and Feasibility of Intervention questionnaires. Items are measured on a 5-point Likert scale (completely disagree to completely agree). Score is calculated mean. An average rating of 4 or higher will be considered feasible/acceptable.
Feasibility of Intervention Questionnaire Ratings | Evaluated at months 2 and 4
  Intervention acceptability and feasibility will be assessed via Acceptability of Intervention and Feasibility of Intervention questionnaires. Items are measured on a 5-point Likert scale (completely disagree to completely agree). Score is calculated mean. An average rating of 4 or higher will be considered feasible/acceptable.
Augmentation Index | Time Frame: Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Augmentation index (a marker for arterial stiffness) will also be assessed using Mobil-O-Graph device.
Biomarkers for Cardiovascular and Metabolic Health - glucose | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up
  Fasting blood will be drawn from the antecubital vein by a trained phlebotomist. Glucose will be measured.
Biomarkers for Cardiovascular and Metabolic Health - HbA1c | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up.
  Fasting blood will be drawn from the antecubital vein by a trained phlebotomist. HbA1c will be measured.
Biomarkers for Cardiovascular and Metabolic Health - c-peptide | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up.
  Fasting blood will be drawn from the antecubital vein by a trained phlebotomist. C-peptide (biomarkers of glycemic control and insulin resistance) will be measured.
Biomarkers for Cardiovascular and Metabolic Health - c-reactive protein | Evaluated at week 1 for baseline, week 16 for post-intervention assessment, and week 32 for follow-up.
  Fasting blood will be drawn from the antecubital vein by a trained phlebotomist. C-reactive protein (CRP; biomarker of system inflammation) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Yan H, Gonzalo-Encabo P, Wilson RL, Christopher CN, Cannon JD, Kang DW, Gardiner J, Perez M, Norris MK, Gundersen D, Hayman LL, Freedman RA, Rebbeck TR, Shi L, Dieli-Conwright CM. Testing home-based exercise strategies in underserved minority cancer patients undergoing chemotherapy (THRIVE) trial: a study protocol. Front Oncol. 2024 Sep 16;14:1427046. doi: 10.3389/fonc.2024.1427046. eCollection 2024. PMID 39351353